CLINICAL TRIAL: NCT04367168
Title: Double-blind, Placebo-controlled Clinical Trial of the Use of Colchicine for the Management of Patients With Mild and Severe SARS-Cov2 Infection
Brief Title: Colchicine in Patients With Mild and Severe Coronavirus Disease
Acronym: ColchiVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The intervention was not effective for the outcomes
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 337420-21-1
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2021-08

CONDITIONS: COVID
Keywords: Colchicine; Coronavirus; Inflammation; Cytokine storm; Clots
MeSH Terms: conditions — Coronavirus Infections; Inflammation; Cytokine Release Syndrome | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled clinical trial to test the security and efficacy of colchicine at a dose of 1.5 mg PO at day 1 followed by 0.5 mg PO BID to complete 10 days of treatment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): Colchicine PO
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo PO
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Colchicine — Colchicine 1mg, 1 ½ pill in day 1 and ½ pill BID during 10 days in both mild and severe COVID-19
  Other Names: Perrigo
  Arms: Colchicine
Drug: Placebo oral tablet — Placebo, 1 ½ pill in day 1 and ½ pill BID during 10 days in both mild and severe COVID-19
  Other Names: Armstrong
  Arms: Placebo

SUMMARY:
The world is currently facing a pandemic due to the outbreak of a new coronavirus causing acute respiratory failure called SARS-Cov2. The majority of patients (8 out of 10) are known to have mild disease, manifested by respiratory tract symptoms associated with fever, headache, and body pain. However, it is possible that the disease progresses to a severe stage, whith the need for mechanical ventilation support associated with high morbidity and mortality. The progression of the disease is mainly due to the appearance of uncontrolled inflammation that also favors the development of disseminated clots. So far, there is no effective treatment to combat coronavirus; however, the use of anti-inflammatory drugs is potentially effective in preventing complications from the disease. In this regard, low dose colchicine is relatively safe and effective as an anti-inflammatory. It has been used for many years in the control of inflammation secondary to the accumulation of uric acid crystals. The aim of this study is to test if the administration of colchicine at a dose of 1.5 mg the first day and subsequently 0.5 mg BID until completing 10 days of treatment is effective as a treatment for inflammation related symptoms in patients with mild and severe disease secondary to coronavirus infection. The primary outcome is improvement of symptoms related to inflammation and avoiding progression to severe and critical stages of the disease. Colchicine can be discontinued before the end of 10 days in case of serious adverse effects or if the patient progresses to the critical stages of the disease.

DETAILED DESCRIPTION:
This a placebo-controlled double-blind clinical trial to test the efficacy and security of colchicine 1.5 mg at day one followed by 0.5 mg BID to complete 10 days of treatment. The researchers will recruit patients 18-70 years of age who are hospitalized because of the diagnosis of mild or severe COVID-19. Patients will be randomized to receive one of the treatment arms, colchicine or placebo. The aim of the study is to evaluate if colchicine may be able to improve the outcomes in patients with mild and severe COVID-19. Patients will be followed-up during the entire hospitalization time and during convalescence. The importance of this intervention is highlighted because currently, there is not an effective treatment for the virus, nor for the prevention of the cytokine storm or the disseminated intravascular coagulation. Therefore, an early intervention to prevent the development of these complications would be valuable to prevent the morbi-morbidity secondary to severe and critical COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Diagnosed with COVID-19 with mild or severe disease
3. Who must receive in-hospital care at the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
4. Who are able to take pills PO

Exclusion Criteria:

* 1. Concomitant participation in another clinical trial. 2. Hypersensitivity to colchicine 3. Pregnancy and lactation 4. Over 70 years 5. Kidney failure with creatinine clearance <30 mL / min. 6. Known liver failure 7. Concomitant medication that has interactions with colchicine and that due to its indication cannot be suspended or substituted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with improvement in body temperature, myalgia, arthralgia, total lymphocyte count, D-dimer, fibrinogen and ferritin levels | Up to 24 days
  Resolution of fever, myalgia and arthralgia and 50% improvement of total lymphocyte count, D-dimer, fibrinogen and ferritin
Progression to severe disease | Up to 10 days
  At least one of the following: respiratory failure, respiratory rate > 30 rpm, oxygen saturation < 92%, PaO2/FiO2 < 300 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: José J Torres-Ruiz, MD, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of the clinical trial
Access Criteria: Reviewers of scientific journals and researchers who contact the principal researcher by e-mail

REFERENCES:
- [Derived] Absalon-Aguilar A, Rull-Gabayet M, Perez-Fragoso A, Mejia-Dominguez NR, Nunez-Alvarez C, Kershenobich-Stalnikowitz D, Sifuentes-Osornio J, Ponce-de-Leon A, Gonzalez-Lara F, Martin-Nares E, Montesinos-Ramirez S, Ramirez-Alemon M, Ramirez-Rangel P, Marquez MF, Plata-Corona JC, Juarez-Vega G, Gomez-Martin D, Torres-Ruiz J. Colchicine Is Safe Though Ineffective in the Treatment of Severe COVID-19: a Randomized Clinical Trial (COLCHIVID). J Gen Intern Med. 2022 Jan;37(1):4-14. doi: 10.1007/s11606-021-07203-8. Epub 2021 Nov 9. PMID 34755269